CLINICAL TRIAL: NCT06254872
Title: Qoyangnuptu: Peer Mentor Pilot 1
Brief Title: Qoyangnuptu: Peer Mentor
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Arizona University (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2125144
Record Dates: First submitted 2024-01-29; First posted 2024-02-12 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-08

CONDITIONS: Mental Health Wellness 1
Keywords: American Indian / Alaska Native; peer mentor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Peer Mentors (Experimental): Participants will be trained in how to be peer mentors to anonymous participants through a smartphone app. Participants will provide daily prompts to their mentees to encourage anonymous discussion in the group chat feature of the smartphone app. Participants will provide daily encouragement to their mentees to use features of the smartphone app to practice mindfulness skills.
  Interventions: Behavioral: Peer Mentors

INTERVENTIONS:
Behavioral: Peer Mentors — Peer mentors provide daily guidance and encouragement to mentees via smartphone app based on training.
  Other Names: Sunrise Peer Mentors

SUMMARY:
The goal of this clinical trial is to learn about the impacts of participating in a peer mentor program in a Southwestern Tribal Community. The main questions it aims to answer are:

* In American Indian/Alaska Native communities with unique cultural characteristics, how should a youth-focused sociotechnical behavioral health intervention be designed to encourage sustained engagement and positively impact indicators of behavioral health?;
* How can interactive technical interventions be designed to best support sustained community engagement in a challenged network environment?

Participants will:

* Be trained as peer mentors
* Be trained in how to use the QI App to communicate with mentees
* Guide daily conversation prompts with a group of 3 mentees via the QI App
* Provide daily encouragement to mentees to engage with mindfulness activities on the QI App

ELIGIBILITY:
Inclusion Criteria:

* Member of Southwestern Tribal Community
* Has a smartphone
* Has access to the Internet with the smartphone at least once per day

Exclusion Criteria:

* Has not completed GED/High School Diploma

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
To measure the acceptability of the Peer Mentorship Program | Baseline, 6 weeks after starting as a mentor, 12 weeks after starting as a mentor
  Through qualitative interviews, the investigators will determine the acceptability of the Peer Mentorship Program. 4 participants will be interviewed after they have participated in the Peer Mentorship Program as Peer Mentors for 6 weeks.

SECONDARY OUTCOMES:
Impact of participation in Peer Mentorship Program as Peer Mentor on attitudes towards seeking professional mental health assistance. | Baseline, 6 weeks after starting as a mentor, 12 weeks after starting as a mentor
  Measured by the Attitudes Towards Seeking Professional Psychological Help - Short Form Scale before participating as a Peer Mentor, 6 weeks into participating as a Peer Mentor, and 12 weeks after starting as a peer mentor.
  The Attitudes Towards Seeking Professional Psychological Help is a 10-item measure used to assess attitudes towards seeking professional psychological help on a 4-point Likert scale, ranging from 0 to 3. Higher total score indicates more positive attitudes towards seeking seeking professional psychological help and is associated with lower levels of stigma against mental illness.
Impact of participation in Peer Mentorship Program as Peer Mentor on measures of depression. | Baseline, 6 weeks after starting as a mentor, 12 weeks after starting as a mentor
  Patient Health Questionnaire-9 before participating as a Peer Mentor, 6 weeks into participation as a Peer Mentor, and 12 weeks after starting as a peer mentor.
  The Patient Health Questionnaire-9 is a 9-item measure used to assess frequency that a participant experiences depressive symptoms. Each item is score on a 4-point scale from 0 ("not at all") to 3 ("every day"). Higher total scores indicate more frequent experience of depressive symptoms.
Impact of participation in Peer Mentorship Program as Peer Mentor on measures of stress. | Baseline, 6 weeks after starting as a mentor, 12 weeks after starting as a mentor
  Perceived Stress Scale 4 before participating as a Peer Mentor, 6 weeks into participation as a Peer Mentor, and 12 weeks after starting as a peer mentor.
  The Perceived Stress Scale 4 measures participant perceptions of their thoughts and feelings over the past month on 4 items. Each item is scored on a 5-point scale from from 0 ("Never") to 4 ("Very Often"). Higher scores indicate higher levels of stress.
Impact of participation in Peer Mentorship Program as Peer Mentor on measures of mindfulness. | Baseline, 6 weeks after starting as a mentor, 12 weeks after starting as a mentor
  State Mindfulness Scale Physical Activity before participating as a Peer Mentor, 6 weeks into participation as a Peer Mentor, and 12 weeks after starting as a peer mentor.
  The State Mindfulness Physical Activity scale is a 12 item measure with six items assessing state mindfulness of the mind (i.e., thoughts and emotions) and six items assessing state mindfulness of the body (i.e., movement, body sensations, muscle engagement). The response scale is 0 - 4, with anchors of Not at all (0) and Very much (4). Initial evidence supports a bi-factor structure of the measure in which both a general state mindfulness factor and two specific factors (mind and body) are supported. The bi-factor structure supports the use of using a single score to capture overall state mindfulness, but also the use of two scores capture mindfulness of the mind and mindfulness of the body.
Impact of participation in Peer Mentorship Program as Peer Mentor on measures of quiet ego. | Baseline, 6 weeks after starting as a mentor, 12 weeks after starting as a mentor
  Quiet Ego Scale before participating as a Peer Mentor, 6 weeks into participation as a Peer Mentor, and 12 weeks after starting as a peer mentor.
  The Quiet Ego Scale is a 14 item measure that assesses detached awareness, inclusive identity, perspective taking, and growth. Each item is assessed on a 5-point Likert scale from 1 ("strongly disagree") to 5 ("strongly agree"). A higher score indicates a stronger quiet ego.
Impact of participation in Peer Mentorship Program as Peer Mentor on measures of social connectedness. | Baseline, 6 weeks after starting as a mentor, 12 weeks after starting as a mentor
  University of California Los Angeles Loneliness Scale 3 before participating as a Peer Mentor, 6 weeks into participation as a Peer Mentor, and 12 weeks after starting as a peer mentor.
  The Loneliness Scale 3 comprises 3 questions that measure 3 dimensions of loneliness: relational connectedness, social connectedness, and self-perceived isolation. Each item is measured on a 3-point scale from 1 ("Hardly Ever") to 3 ("Often"). Higher scores indicate greater perceptions of loneliness.

CONTACTS AND LOCATIONS:
Overall Officials: Morgan Vigil-Hayes, PhD, Principal Investigator — Northern Arizona University
Locations (1):
- Northern Arizona University, Flagstaff, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
Individual participants will be from a small, rural community and confidentiality can be easily breached if individual participant data is revealed.

REFERENCES:
- [Background] Vigil-Hayes M, Collier AF, Hagemann S, Castillo G, Mikkelson K, Dingman J, Munoz A, Luther J, McLaughlin A. Integrating Cultural Relevance into a Behavioral mHealth Intervention for Native American Youth. Proc ACM Hum Comput Interact. 2021 Apr;5(CSCW1):165. doi: 10.1145/3449239. PMID 34676359
- [Background] Vigil-Hayes M, Futterman Collier A, Castillo G, Blackhorse D, Awbery N, Abrahim JP. Designing a Mobile Game That Develops Emotional Resiliency in Indian Country. Ext Abstr Hum Factors Computing Syst. 2019 May;2019:LBW2122. doi: 10.1145/3290607.3312790. PMID 32455346
- [Background] Picco L, Abdin E, Chong SA, Pang S, Shafie S, Chua BY, Vaingankar JA, Ong LP, Tay J, Subramaniam M. Attitudes Toward Seeking Professional Psychological Help: Factor Structure and Socio-Demographic Predictors. Front Psychol. 2016 Apr 25;7:547. doi: 10.3389/fpsyg.2016.00547. eCollection 2016. PMID 27199794
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Cox AE, Ullrich-French S, Howe HS, Cole AN. A pilot yoga physical education curriculum to promote positive body image. Body Image. 2017 Dec;23:1-8. doi: 10.1016/j.bodyim.2017.07.007. Epub 2017 Aug 14. PMID 28818786
- [Background] Hughes ME, Waite LJ, Hawkley LC, Cacioppo JT. A Short Scale for Measuring Loneliness in Large Surveys: Results From Two Population-Based Studies. Res Aging. 2004;26(6):655-672. doi: 10.1177/0164027504268574. PMID 18504506
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941